CLINICAL TRIAL: NCT01093222
Title: Phase II Study of Sorafenib (NSC-724772) and Erlotinib (NSC-718781) in Patients With Advanced Gallbladder Carcinoma or Cholangiocarcinoma
Brief Title: Sorafenib Tosylate and Erlotinib Hydrochloride in Treating Patients With Locally Advanced, Unresectable, or Metastatic Gallbladder Cancer or Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02027; NCI-2011-02027 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0941; CDR0000668246; S0941 (Other: SWOG); S0941 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-03

CONDITIONS: Extrahepatic Bile Duct Adenocarcinoma; Gallbladder Adenocarcinoma; Gallbladder Adenocarcinoma With Squamous Metaplasia; Hilar Cholangiocarcinoma; Recurrent Extrahepatic Bile Duct Carcinoma; Recurrent Gallbladder Carcinoma; Undifferentiated Gallbladder Carcinoma; Unresectable Extrahepatic Bile Duct Carcinoma; Unresectable Gallbladder Carcinoma
MeSH Terms: conditions — Klatskin Tumor; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Erlotinib Hydrochloride; Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate and erlotinib hydrochloride) (Experimental): Patients receive sorafenib tosylate PO twice daily and erlotinib hydrochloride PO once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib Hydrochloride; Drug: Sorafenib Tosylate

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase II trial is studying how well giving sorafenib tosylate together with erlotinib hydrochloride works in treating patients with locally advanced, unresectable, or metastatic gallbladder cancer or cholangiocarcinoma. Sorafenib tosylate and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess the progression-free survival in patients with unresectable or metastatic gallbladder carcinoma or cholangiocarcinoma treated with the combination of sorafenib (sorafenib tosylate) and erlotinib (erlotinib hydrochloride).

II. To assess the overall survival in patients with unresectable or metastatic gallbladder carcinoma or cholangiocarcinoma treated with the combination of sorafenib and erlotinib.

III. To assess the objective response rate. IV. To assess the frequency and severity of toxicities. V. To collect specimens for banking for future research.

OUTLINE: This is a multicenter study.

Patients receive sorafenib tosylate orally (PO) twice daily and erlotinib hydrochloride PO once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or pathologically confirmed gallbladder carcinoma or cholangiocarcinoma

  * No ampullary carcinoma
* Locally advanced unresectable or distant metastatic disease
* Measurable disease
* Patients with biliary obstruction must have decompression of the biliary tree by ERCP and stenting or percutaneous drainage
* No prior systemic treatment for metastatic or unresectable locally advanced disease
* No known brain metastases
* Zubrod performance status of 0-1
* Leukocyte count ≥ 3,000/mm^3
* ANC ≥ 1,000/mm^3
* Platelet count ≥100,000/mm^3
* Total serum bilirubin ≤ 1.5 times upper limit of normal (ULN)

  * For patient who had decompression of the biliary tree within the past 14 days, stability of the bilirubin level needs to be confirmed with two measurements within 5 to 7 days of each other
* Serum albumin ≥ 2.5 g/dL
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN for liver metastases)
* Creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Fertile patients must agree to use effective contraception
* No active biliary sepsis
* No bleeding diathesis
* No uncontrolled or clinically significant cardiovascular disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * Uncontrolled angina within the past 6 months
  * NYHA class II-IV congestive heart failure
  * Grade 3 cardiac valve dysfunction
  * Cardiac arrhythmia not controlled by medication
  * History of stroke or transient ischemic attack within the past 6 months
  * History of arterial thrombotic event of any type in the past 6 months
* No uncontrolled hypertension, as evidenced by systolic BP ≥ 150 mm Hg or diastolic BP ≥ 100 mm Hg, within the past 28 days
* Must be able to swallow and tolerate oral medications

  * No gastrointestinal tract disease or prior abdominal surgery that results in an inability to absorb oral medication
* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free within the past 3 years
* No concurrent grapefruit or its juice
* At least 6 months since 1 adjuvant or neoadjuvant regimen of chemotherapy, hormonal therapy, immunotherapy, radiotherapy (to < 25% of bone marrow only), or chemoradiotherapy before documented recurrence or metastatic disease
* No prior treatment with any antiangiogenic agent or any EGFR inhibitors for any reason
* Concurrent multiple anti-hypertensive medications allowed
* No plans to receive concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or any other therapy, including herbal or alternative medications for treatment of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2012-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, Principal Investigator — SWOG Cancer Research Network
Locations (141):
- United States (141):
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Sutter Cancer Research Consortium, Novato, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Central Illinois CCOP, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Boston Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib and Erlotinib: Patients receive sorafenib tosylate 400 mg PO twice daily and erlotinib hydrochloride 100 mg PO once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Sorafenib and Erlotinib
Started | 40
Eligible and Began Protocol Therapy | 34
Completed | 0
Not Completed | 40
Not completed — Ineligible | 6
Not completed — Adverse Event | 7
Not completed — Progression/relapse | 24
Not completed — Death | 2
Not completed — Not protocol specified | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy
Arm/Group | Sorafenib and Erlotinib
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 63 [49 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Zubrod Performance Status [Number; unit: participants] — Zubrod Performance Status Scale: 0 - Fully active, able to carry on all pre-disease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light sedentary nature; 2 - Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours; 3 - Capable of limited self-care, confined to bed or chair more than 50% of waking hours; 4 - Completely disabled, cannot carry on any self-care, totally confined to bed or chair
  participants
    0 | 19
    1 | 15
Chemotherapy, multiple agents [Number; unit: participants]
  Yes | 1
  No | 33
Prior Surgery [Number; unit: participants]
  Yes | 14
  No | 20
Current Status of Disease [Number; unit: participants]
  Distant Metastatic | 28
  Locally Advanced | 6
Primary Cancer [Number; unit: participants]
  Cholangiocarcinoma | 20
  Gallbladder | 14
Prior Radiation Therapy [Number; unit: participants]
  Yes | 0
  No | 34
Setting of Prior Chemotherapy [Number; unit: participants]
  Adjuvant | 1
  Neoadjuvant | 0
  None | 33

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 3 years
Population: Eligible patients who began protocol therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib and Erlotinib
Number analyzed (Participants) | 34
months | 6 [3 to 8]

2. Primary Outcome: Progression-free Survival
Description: From date of registration to date of first documentation of progression or symptomatic deterioration (as defined in protocol), or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact.
Time Frame: Up to 3 years
Population: Eligible patients who began protocol therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib and Erlotinib
Number analyzed (Participants) | 34
months | 2 [2 to 3]

3. Secondary Outcome: Objective Response
Description: Complete response (CR) is complete disappearance of all target and non-target lesions, no new lesions and no disease related symptoms. Partial response (PR) is a greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. Confirmed response is two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. Partial response is two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration. Unconfirmed CR is one objective status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR. Unconfirmed PR is one objective status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Up to 3 years
Population: Eligible patients who began protocol therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib and Erlotinib
Number analyzed (Participants) | 34
percentage of participants | 6 [1 to 20]

4. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 3 years
Population: Eligible patients who received any treatment and were assessed for toxicity were included in the adverse event summaries. Any CTCAE v4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Sorafenib and Erlotinib
Number analyzed (Participants) | 34
Participants
  Abdominal pain | 1
  Alanine aminotransferase increased | 4
  Alkaline phosphatase increased | 3
  Allergic reaction | 1
  Aspartate aminotransferase increased | 3
  Blood bilirubin increased | 2
  Death NOS | 1
  Dehydration | 1
  Diarrhea | 3
  Erythema multiforme | 1
  Fatigue | 1
  Gastric perforation | 1
  Hepatic failure | 1
  Hepatic infection | 1
  Hepatic necrosis | 1
  Hypertension | 5
  Hypoalbuminemia | 1
  Hypokalemia | 2
  Hypophosphatemia | 3
  Hypoxia | 1
  Lymphocyte count decreased | 1
  Mucositis oral | 1
  Nausea | 1
  Pain | 1
  Palmar-plantar erythrodysesthesia syndrome | 2
  Platelet count decreased | 1
  Rash acneiform | 1
  Rash maculo-papular | 1
  Thromboembolic event | 1

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Sorafenib and Erlotinib
Serious Adverse Events (participants affected / at risk) | 17/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib and Erlotinib (N=34)
Cardiac arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 6
Multi-organ failure (General disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1
Hepatic necrosis (Hepatobiliary disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Device related infection (Infections and infestations) | 1
Hepatic infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib and Erlotinib (N=34)
Anemia (Blood and lymphatic system disorders) | 11
Leukocytosis (Blood and lymphatic system disorders) | 2
Conjunctivitis (Eye disorders) | 2
Dry eye (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 20
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 17
Oral pain (Gastrointestinal disorders) | 3
Rectal hemorrhage (Gastrointestinal disorders) | 3
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 2
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 17
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 2
Pain (General disorders) | 6
Urinary tract infection (Infections and infestations) | 3
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 18
Alkaline phosphatase increased (Investigations) | 17
Aspartate aminotransferase increased (Investigations) | 22
Blood bilirubin increased (Investigations) | 12
Creatinine increased (Investigations) | 2
INR increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 10
Weight loss (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 3
Dysarthria (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 5
Urine discoloration (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 12
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
The first stage of accrual was met with 40 registered patients. Insufficient number of patients were alive and free from progression at four months to warrant accruing to a second stage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less